CLINICAL TRIAL: NCT04689828
Title: PSMAfore: A Phase III, Open-label, Multi-Center, Randomized Study Comparing 177Lu-PSMA-617 vs. a Change of Androgen Receptor-Directed Therapy in the Treatment of Taxane Naïve Men With Progressive Metastatic Castrate Resistant Prostate Cancer
Brief Title: 177Lu-PSMA-617 vs. Androgen Receptor-Directed Therapy in the Treatment of Progressive Metastatic Castrate Resistant Prostate Cancer
Acronym: PSMAfore
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAA617B12302; 2023-507772-50-00 (Other: EU CTIS)
Record Dates: First submitted 2020-12-09; First posted 2020-12-30 (Actual); Results first posted 2025-10-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms
Keywords: 177Lu-PSMA-617; Androgen receptor-directed therapy; ARDT; Metastatic castrate resistant prostate cancer; mCRPC; Radiographic progression free survival; rPFS; Castrate resistant prostate cancer; CRPC; Prostate-specific membrane antigen; PSMA
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto; gallium 68 PSMA-11

STUDY DESIGN:
Intervention Model Description: Patients randomized to ARDT treatment had an option to crossover to 177Lu-PSMA-617 treatment after central confirmation of radiographic progression.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 177Lu-PSMA-617 (Experimental): Participants received 7.4 GBq (200 mCi) +/- 10% 177Lu-PSMA-617 once every 6 weeks for 6 cycles. Best supportive care, including ADT could be used.
  Interventions: Drug: 177Lu-PSMA-617; Drug: 68Ga-PSMA-11
- Androgen receptor-directed therapy (ARDT) (Active Comparator): For participants randomized to the ARDT arm, abiraterone or enzalutamide was administered per the physician's orders. Best supportive care, including Androgen deprivation therapy (ADT) could be used.
  Interventions: Drug: 68Ga-PSMA-11; Drug: ARDT

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — administered intravenously once every 6 weeks (1 cycle) for 6 cycles
  Arms: 177Lu-PSMA-617
Drug: 68Ga-PSMA-11 — single intravenous dose of approximately 150 MBq. Administered dose must not be lower than 111 MBq or higher than 185 MBq (3 - 5 mCi).
Drug: ARDT — administered orally on a continuous basis, as per package insert and guidelines
  Other Names: Comparator
  Arms: Androgen receptor-directed therapy (ARDT)

SUMMARY:
The purpose of this study is to determine whether 177Lu-PSMA-617 improves the Radiographic progression-free survival (rPFS) or Overall Survival (OS) compared to a change in Androgen receptor-directed therapy (ARDT) in metastatic castrate resistant prostate cancer (mCRPC) participants that were previously treated with an alternate ARDT and not exposed to a taxane-containing regimen in the CRPC or mHSPC settings.

469 participants were randomized (235 in the 177Lu-PSMA-617 group and 234 in the ARDT group.

DETAILED DESCRIPTION:
This is a phase III, open label, multicenter randomized study evaluating the superiority of 177Lu-PSMA-617 over a change of ARDT treatment in prolonging rPFS. The primary endpoint of rPFS is to assess via blinded independent centralized review (BICR) of radiographic images provided by the treating physician and as outlined in PCWG3 modified RECIST v 1.1 Guidelines.

The study also evaluates whether 177Lu-PSMA-617 improves the overall survival (OS) in participants with progressive PSMA-positive mCRPC compared to participants treated with a change in ARDT treatment. OS is defined as the time from randomization to death due to any cause.

Treatment duration: approximately 43 months.

Screening period At screening, the participants are assessed for eligibility and undergo a 68Ga-PSMA-11 positron emission tomography (PET)/computed tomography (CT) scan to evaluate PSMA positivity. Only participants with PSMA positive cancer and confirmed eligibility criteria are randomized.

Randomization period The participants are randomized 1:1 to receive 177Lu-PSMA-617 or a change of the ARDT treatment. The ARDT change includes approved Androgen Receptor (AR) axis targeted therapy (abiraterone or enzalutamide). Supportive care is allowed in both arms at the discretion of the investigator and includes available care for the eligible participant according to best institutional practice for mCRPC treatment, including androgen deprivation therapy (ADT). Investigational agents, biological products, immunotherapy, cytotoxic chemotherapy, other systemic radioisotopes (e.g. radium-223), poly (adenosine diphosphate-ribose) polymerase (PARP) inhibitors or hemi-body radiotherapy treatment is not to be administered during the study treatment period. ARDT is not to be administered concomitantly with 177Lu-PSMA-617. After implementation of Protocol Amendment v4, crossover will be allowed regardless of radiographic progression.

Treatment period • 177Lu-PSMA-617 treatment arm Participants randomized to the investigational arm receive 7.4 GBq +/- 10% of 177Lu-PSMA-617 once every 6 weeks for 6 cycles. Best supportive care, including ADT, could be used.

After the last day of study treatment, the participants have to have an End of Treatment (EOT) visit and enter the Post-treatment Follow-up.

• ARDT treatment arm For participants randomized to the ARDT treatment arm, the change of ARDT treatment for each participant is selected by the treating physician prior to randomization and is administered per the physician's orders. Best supportive care, including ADT, could be used. After, the participants have to have an End of Treatment (EOT) and enter the Post-treatment Follow-up.

In absence of safety concerns, every effort should be made to keep the participant on the randomized treatment until BICR-determined radiographic progression (up to implementation of Protocol Amendment v4).

End of Treatment

Randomized treatment may be discontinued if:

* The participant, sponsor or investigator chooses to discontinue treatment
* Toxicity
* Completion of the 6 cycles of 177Lu-PSMA-617
* Serious non-compliance to the protocol
* Disease progression (determined by BICR up to implementation of Protocol Amendment v4)
* Upon implementation of Protocol Amendment v4, participants with ongoing treatment with ARDT will discontinue study drug and either crossover or receive SOC per their treating physician off trial PSA progression is strongly discouraged as a criterion for initiation of a new neoplastic therapy prior to BICR-determined progression. PCWG3 guidelines should be followed to guide discontinuation of treatment End of Treatment visit must be performed ≤ 7 days after the last day of study treatment period. EOT is to occur before the participant ienters the post-treatment Follow-up period of the study and before the initiation of any subsequent anticancer treatment, .

If a participant withdraws consent for the treatment period of the study, an EOT must be done and the participant will enter the Post-treatment Follow-up unless he specifically withdraws post-treatment Follow-up.

Crossover period Upon confirmation of rPFS by BICR, participants randomized to the ARDT arm could either be allowed to crossover to receive 177Lu-PSMA-617 within 28 days of central confirmation of radiographic progression or could continue to receive any other therapy per the discretion of the treating physician in the Post-treatment Follow-up.

In order for a participant randomized to the ARDT arm to cross over to receive 177Lu-PSMA-617, he must meet the following criteria:

* Confirmed radiographical progression as assessed by BICR. (After implementation of Protocol Amendment v4, radiographic progression is not required.)
* No intervening antineoplastic therapy is administered after the randomized treatment
* Any unresolved toxicity from prior therapy has to be controlled and can be no greater than CTCAE grade 2 or baseline at the time of registration for crossover.
* ECOG performance status 0-1 at the time of registration for crossover
* Adequate organ function at the time of registration for crossover
* Agreement to continue with the study visit schedule

A participant, who is deemed to have disease progression per investigator assessment, but not by BICR, is not eligible to cross over at that time. Such participant should continue to receive randomized study treatment until progression determined by BICR up to implementation of Protocol Amendment v4.

If crossover to 177Lu-PSMA-617 is selected, then 177Lu-PSMA-617 will be administered with the same dose/schedule as for participants who were initially randomized to receive 177Lu-PSMA-617 as described above.

After the last day of study treatment period of 177Lu-PSMA-617 or upon second radiographic progression (rPFS2), the participants must have a second End of Treatment (EOT2) visit performed ≤ 7 days and enter the Post-treatment Follow-up. The participant can receive any other therapy per the discretion of the treating physician in the Post-treatment Follow-up.

Post-treatment Follow-up period:

* 30-day Safety Follow-up: All randomized and/or treated participants are to have a safety follow-up conducted approximately 30 days after the EOT visit.
* Long term follow-up:

Long term follow-up starts after the 30 Days Safety follow-up and lasts until the patient expires, is lost to follow-up or withdraws consent.

In long term follow-up safety and efficacy information is collected:

* Safety: all medically significant adverse events (all SAEs) deemed to be related to 177Lu-PSMA-617. This includes potential late onset radiation toxicity. For participants who receive 177Lu-PSMA-617 in the 177Lu-PSMA-617 arm or in crossover, the following adverse events is captured beyond the 30 day safety period regardless of relationship to study treatment and whether new anticancer therapy has been initiated: hematologic toxicities with primary focus on myelosuppression and thrombocytopenia (including need for transfusion or use of growth factors), renal failure, xerostomia, xerophthalmia, secondary malignancies. After implementation of Protocol Amendment v4, 177Lu-PSMA-617 exposed participants will be discontinued from the trial once enrolled in the Long-term Safety study.
* Efficacy: Tumor assessments must be performed every 8 weeks after first dose of study treatment for the first 24 weeks (week 9, 17, 25) and then every 12 weeks (week 37, 49, etc.) until confirmation of radiographic progression by BICR regardless of whether treatment has been discontinued or new anticancer therapy initiated. After implementation of Protocol Amendment v4, tumor assessments need to continue only for patients actively treated with 177Lu-PSMA-617 as crossover therapy.

The long-term follow-up period also includes the collection of survival information and other assessments.

Other: Other data collected during long-term follow-up includes short physical exam, blood sampling for hematology, chemistry testing, coagulation, DNA and tumor samples for biomarkers. The visits are carried out every 12 weeks (± 28 days) .

Participants who receive 177Lu-PSMA-617 and remain in follow-up on the trial at the sponsor's completion of the study will be asked to join a separate study of long-term safety for a duration of up to 10 years from start of 177Lu-PSMA-617 treatment.

If the participant withdraws consent for the collection of blood samples, PROs, and imaging assessments during the long-term follow-up, information on survival subsequent therapy, and related SAEs is collected.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Participants must be adults >= 18 years of age.
* Participants must have an ECOG performance status of 0 to 1.
* Participants must have histological pathological, and/or cytological confirmation of adenocarcinoma of the prostate.
* Participants must be 68Ga-PSMA-11 PET/CT scan positive, and eligible as determined by the sponsor's central reader.
* Participants must have a castrate level of serum/plasma testosterone (< 50 ng/dL or < 1.7 nmol/L).
* Participants must have progressed only once on prior second generation ARDT (abiraterone, enzalutamide, darolutamide, or apalutamide).

  * First generation androgen receptor inhibitor therapy (e.g. bicalutamide) is allowed but not considered as prior ARDT therapy.
  * Second generation ARDT must be the most recent therapy received.
* Participants must have progressive mCRPC. Documented progressive mCRPC will be based on at least 1 of the following criteria:

  * Serum/plasma PSA progression defined as 2 increases in PSA measured at least 1 week apart. The minimal start value is 2.0 ng/mL; 1.0 ng/mL is the minimal starting value if confirmed rise in PSA is the only indication of progression.
  * Soft-tissue progression defined [PCWG3-modified RECIST v1.1 (Eisenhauer et al 2009, Scher et al 2016)].
  * Progression of bone disease: two new lesions; only positivity on the bone scan defines metastatic disease to bone (PCWG3 criteria (Scher et al 2016)).
* Participants must have >= 1 metastatic lesion that is present on baseline CT, MRI, or bone scan imaging obtained prior to randomization.
* Participants must have recovered to =< Grade 2 from all clinically significant toxicities related to prior therapies (i.e. prior chemotherapy, radiation, etc.) except alopecia.
* 11. Participants must have adequate organ function:

  * Bone marrow reserve:
  * ANC >= 1.5 x 109/L
  * Platelets >= 100 x 109/L
  * Hemoglobin >= 9 g/dL
  * Hepatic:
  * Total bilirubin < 2 x the institutional upper limit of normal (ULN). For participants with known Gilbert's Syndrome =< 3 x ULN is permitted.
  * ALT or AST =< 3.0 x ULN OR =< 5.0 x ULN for participants with liver metastases.
  * Renal:
  * eGFR >= 50 mL/min/1.73m2 using the Modification of Diet in Renal Disease (MDRD) equation.
* Albumin >= 2.5 g/dL. -. Candidates for change in ARDT as assessed by the treating physician: • Participants cannot have previously progressed nor had intolerable toxicity to both enzalutamide and abiraterone.

Exclusion Criteria:

* Previous treatment with any of the following within 6 months of randomization: Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, hemi-body irradiation.
* Previous PSMA-targeted radioligand therapy.
* Prior treatment with cytotoxic chemotherapy for castration resistant or castrate sensitive prostate cancer (e.g., taxanes, platinum, estramustine, vincristine, methotrexate, etc.), immunotherapy or biological therapy [including monoclonal antibodies]. [Note: Taxane exposure (maximum 6 cycles) in the adjuvant or neoadjuvant setting is allowed if 12 months have elapsed since completion of this adjuvant or neoadjuvant therapy. Prior treatment with sipuleucel-T is allowed].
* Any investigational agents within 28 days prior to day of randomization.
* Known hypersensitivity to any of the study treatments or its excipients or to drugs of similar classes.

  -. Concurrent cytotoxic chemotherapy, immunotherapy, radioligand therapy, PARP inhibitor, biological therapy, or investigational therapy.
* Transfusion or use of bone marrow stimulating agents for the sole purpose of making a participant eligible for study inclusion.
* Participants with a history of CNS metastases who are neurologically unstable, symptomatic, or receiving corticosteroids for the purpose of maintaining neurologic integrity. Participants with CNS metastases are eligible if received therapy (surgery, radiotherapy, gamma knife), asymptomatic and neurologically stable without corticosteroids. Participants with epidural disease, canal disease and prior cord involvement are eligible if those areas have been treated, are stable, and not neurologically impaired.
* Symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression.
* History or current diagnosis of the following ECG abnormalities indicating significant risk of safety for study participants:

  * Concomitant clinically significant cardiac arrhythmias, e.g. sustained ventricular tachycardia, complete left bundle branch block, high-grade AV block (e.g., bifascicular block, Mobitz type II and third degree AV block).
  * History of familial long QT syndrome or known family history of Torsades de Pointe.
  * Cardiac or cardiac repolarization abnormality, including any of the following: History of myocardial infarction (MI), angina pectoris, or CABG within 6 months prior to starting study treatment.
* Concurrent serious (as determined by the Principal Investigator) medical conditions, including, but not limited to New York Heart Association class III or IV congestive heart failure, history of congenital prolonged QT syndrome, uncontrolled infection, known active hepatitis B or C or other significant co-morbid conditions that in the opinion of the investigator would impair study participation or cooperation.

  * HIV-infected participants who are at a low risk of AIDS-related outcomes may participate in this trial.
  * Participants with an active documented COVID-19 infection (any grade of disease severity) at time of informed consent may be included only when completely recovered (in accordance with local guidance).
* Diagnosed with other malignancies that are expected to alter life expectancy or may interfere with disease assessment. However, participants with a prior history of malignancy that has been adequately treated and who have been disease free and treatment free for more than 3 years prior to randomization, are eligible, as are participants with adequately treated non-melanoma skin cancer and superficial bladder cancer.
* Sexually active males unwilling to use a condom during intercourse while taking study treatment and for 14 weeks after stopping study treatment. A condom is required for all sexually active male participants to prevent them from fathering a child AND to prevent delivery of study treatment via seminal fluid to their partner.

In addition, male participants must not donate sperm for the time period specified above. If local regulations deviate from the contraception methods listed above to prevent pregnancy, local regulations apply and will be described in the ICF.

* Unmanageable concurrent bladder outflow obstruction or urinary incontinence. Note: Participant with bladder outflow obstruction or urinary incontinence, which is manageable and controlled with best available standard of care (incl. pads, drainage) are allowed.
* History of somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study.
* Any condition that precludes raised arms position.
* Eligible for treatment(s) other than ARDT based on presence of any mutations or biomarkers that are known as predictors of better response (e.g., AR-V7 or BRCA).
* Not able to understand and to comply with study instructions and requirements.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer study.
Enrollment: 469 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-10-02 (Actual); Study Completion 2026-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (65):
- United States (20):
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Tulane Uni Health Sciences Center, New Orleans, Louisiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - WA Uni School Of Med, St Louis, Missouri
  - Urology Cancer Center PC, Omaha, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - NYU Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Ctr, New York, New York
  - Mount Sinai Hosp Med School, New York, New York
  - Duke Univ Medical Center, Durham, North Carolina
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Uni Of TX MD Anderson Cancer Cntr, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virginia Oncology Associates, Norfolk, Virginia
  - Onco Hemato Asso of SW Virginia, Roanoke, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Austria (3):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (4):
  - Novartis Investigative Site, Roeselare, West-Vlaanderen
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Liège
- Canada (2):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Olomouc, Czechia
- France (6):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Villejuif
- Germany (2):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, München
- Netherlands (3):
  - Novartis Investigative Site, Nijmegen, Gelderland
  - Novartis Investigative Site, Maastricht, Limburg
  - Novartis Investigative Site, Utrecht
- Novartis Investigative Site, Gliwice, Silesian Voivodeship, Poland
- Novartis Investigative Site, Bratislava, Slovakia
- Spain (11):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Sweden (3):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
- Switzerland (3):
  - Novartis Investigative Site, Baden
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- United Kingdom (5):
  - Novartis Investigative Site, Guildford, Surrey
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Coventry
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Middlesbrough

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Fizazi K, Morris MJ, Shore ND, Chi KN, Crosby M, de Bono JS, Herrmann K, Roubaud G, Nagarajah J, Fleming M, Lewis B, Nordquist L, Carnahan N, Ghebremariam S, Hertelendi M, Castellano D, Sartor O. Health-related quality of life, pain, and symptomatic skeletal events with [177Lu]Lu-PSMA-617 in patients with progressive metastatic castration-resistant prostate cancer (PSMAfore): an open-label, randomised, phase 3 trial. Lancet Oncol. 2025 Jul;26(7):948-959. doi: 10.1016/S1470-2045(25)00189-5. Epub 2025 May 26. PMID 40441170
- [Derived] Morris MJ, Castellano D, Herrmann K, de Bono JS, Shore ND, Chi KN, Crosby M, Piulats JM, Flechon A, Wei XX, Mahammedi H, Roubaud G, Studentova H, Nagarajah J, Mellado B, Montesa-Pino A, Kpamegan E, Ghebremariam S, Kreisl TN, Wilke C, Lehnhoff K, Sartor O, Fizazi K; PSMAfore Investigators. 177Lu-PSMA-617 versus a change of androgen receptor pathway inhibitor therapy for taxane-naive patients with progressive metastatic castration-resistant prostate cancer (PSMAfore): a phase 3, randomised, controlled trial. Lancet. 2024 Sep 28;404(10459):1227-1239. doi: 10.1016/S0140-6736(24)01653-2. Epub 2024 Sep 15. PMID 39293462

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Informed consent was obtained from all eligible participants who were randomized via Interactive Response Technology (IRT) to one of the arms in a 1:1 ratio: 177Lu-PSMA-617 or Androgen receptor-directed therapy (ARDT).
Pre-assignment Details: During screening, all participants underwent imaging with the investigational product gallium (68Ga) gozetotide for the purpose of determining eligibility.
Groups:
- 177Lu-PSMA-617 (AAA617): Participants received 7.4 GBq (200 mCi) +/- 10% 177Lu-PSMA-617 once every 6 weeks for 6 cycles. Best supportive care, including ADT could be used.
- Androgen Receptor-directed Therapy (ARDT): For participants randomized to the ARDT arm, the change of ARDT treatment was administered per the physician's orders. Best supportive care, including ADT could be used.
Period: Overall Study
Arm/Group | 177Lu-PSMA-617 (AAA617) | Androgen Receptor-directed Therapy (ARDT)
Started | 235 | 234
Participants Treated | 228 | 232
Full Analysis Set (FAS) (The Full Analysis Set (FAS) comprised all participants to whom study treatment was assigned by randomization.) | 234 | 234
Excluded From FAS (Excluded from Full Analysis Set & Safety Set due to protocol deviation (informed consent not obtained per due process)) | 1 | 0
Participants Not Treated | 7 | 2
Discontinued Study Treatment | 96 | 223
Safety Set (The Safety Set included all participants who received at least one dose of study treatment (i.e., at least one dose of (AAA617 or ARPIs) during the randomized part of the protocol.) | 227 | 232
Completed (Completed = Completed treatment) | 131 | 0
Not Completed | 104 | 234
Not completed — Subject decision | 5 | 5
Not completed — Adverse Event | 12 | 12
Not completed — Physician Decision | 24 | 32
Not completed — Progressive disease | 54 | 173
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Treated but excluded from FAS because of protocol deviation | 1 | 0
Not completed — Treatment ongoing at the data cut-off date of 1-Jan-2025 | 0 | 9
Not completed — Participants not treated | 7 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) comprised all participants to whom study treatment was assigned by randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | 177Lu-PSMA-617 (AAA617) | Androgen Receptor-directed Therapy (ARDT) | Total
Number analyzed (Participants) | 234 | 234 | 468
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (8.70) | 71.9 (7.65) | 71.4 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 234 | 234 | 468
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 2 | 3
  Black or African American | 7 | 5 | 12
  White | 212 | 214 | 426
  Unknown | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Progression Free Survival (rPFS)
Description: rPFS is defined as the time to radiographic progression by Prostate cancer working Group 3 (PCWG3)-modified RECIST v1.1 as assessed by Blinded independent central (BICR) review or death.
Time Frame: median FU (randomization to event or censoring) 3.65 months (range 0-12.3)
Population: The Full Analysis Set (FAS) comprised all participants to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 177Lu-PSMA-617 (AAA617) | Androgen Receptor-directed Therapy (ARDT)
Number analyzed (Participants) | 233 | 234
months | 9.30 [6.77 to NA] — NA: not able to calculate the upper bounds of the 95% Confidence Interval due to insufficient number of participants with events | 5.55 [4.04 to 5.95]
Statistical Analysis 1: Comparison: 177Lu-PSMA-617 (AAA617) vs Androgen Receptor-directed Therapy (ARDT); Test type: Superiority; p = 0.00000001, Log Rank; Stratified; Hazard Ratio (HR) = 0.41, 95% CI 2-sided [0.29 to 0.56]

2. Secondary Outcome: Overall Survival (OS) (Key Secondary Endpoint)
Description: OS is defined as time to death for any cause.
Time Frame: approx. 26.9 months from randomization to cut-off
Population: FAS comprised all participants to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 177Lu-PSMA-617 (AAA617) | Androgen Receptor-directed Therapy (ARDT)
Number analyzed (Participants) | 234 | 234
months | 24.48 [19.55 to 28.94] | 23.13 [19.61 to 25.53]
Statistical Analysis 1: Comparison: 177Lu-PSMA-617 (AAA617) vs Androgen Receptor-directed Therapy (ARDT); Test type: Superiority; p = 0.20, stratified Cox PH model; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.72 to 1.14]

3. Secondary Outcome: Radiographic Progression Free Survival 2 (rPFS2) by Blinded Independent Central Review (BICR)
Description: rPFS2 by BICR is defined as time from the date of crossover (ARDT to 177Lu-PSMA-617) to the date of radiographic disease progression by BICR or death from any cause for participants who crossover from ARDT arm to Lu-PSMA treatment.
Time Frame: From date of crossover until second radiographic progression or death, whichever comes first, assessed up to approx. 32 months
Reporting Status: Not Posted, anticipated posting 2026-09

4. Secondary Outcome: Progression Free Survival (PFS) by Investigator's Assessment
Description: PFS is defined as time from date of randomization to the first documented progression by investigator's assessment (radiographic, clinical, or PSA progression) or death from any cause, whichever occurs first
Time Frame: From date of randomization until date of progression or date of death from any cause, whichever comes first, assessed upFrom date of randomization until date of death from any cause, assessed up to approx. 32 months
Reporting Status: Not Posted, anticipated posting 2026-09

5. Secondary Outcome: Second Progression Free Survival (PFS2) by Investigator's Assessment
Description: PFS2 defined as time from date of randomization to the first documented progression by investigator's assessment (radiographic progression, clinical progression, PSA progression) or death from any cause, whichever occurs first, on next-line of therapy. Next-line therapy was defined as the first new (systemic) anti-neoplastic therapy initiated after discontinuation of study treatment regardless of end of treatment (EoT) reason.
Time Frame: From date of randomization until date of second progression or date of death from any cause, whichever comes first, assessed up to approx. 32 months
Reporting Status: Not Posted, anticipated posting 2026-09

6. Secondary Outcome: PSA50 Response
Description: PSA50 response was defined as the percentage of participants who achieved a ≥ 50% decrease from baseline that is confirmed by a second Prostate specific antigen (PSA) measurement ≥ 4 weeks.
Time Frame: Weeks 12, 24, 48 and anytime during randomized phase
Reporting Status: Not Posted, anticipated posting 2026-09

7. Secondary Outcome: Time to First Symptomatic Skeletal Event (TTSE)
Description: Time to SSE (TTSSE) defined as date of randomization to the date of first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, requirement for radiation therapy to relieve bone pain or death from any cause, whichever occurs first
Time Frame: From date of randomization till EOT or death, whichever happens first, assessed up to approx. 32 months
Reporting Status: Not Posted, anticipated posting 2026-09

8. Secondary Outcome: Time to Radiographic Soft Tissue Progression (TTSTP) Per BICR
Description: TTSTP defined as time from randomization to radiographic soft tissue progression per Prostate cancer working Group 3 (PCWG3)-modified RECIST v1.1 (Soft Tissue Rules of Prostate Cancer Working Group modified Response Evaluation Criteria in Solid Tumors Version 1.1) as assessed by Blinded Independent Central Review (BICR).
Time Frame: From date of randomization until date of soft tissue radiographic progression or date of death from any cause, whichever comes first, assessed up to approx. 32 months
Reporting Status: Not Posted, anticipated posting 2026-09

9. Secondary Outcome: Time to Chemotherapy (TTCT)
Description: TTCT defined as time from randomization to initiation of the first subsequent chemotherapy or death, whichever occurs first. Since participants in ARPI arm were allowed to crossover to [177Lu]Lu-PSMA-617 (AAA617) arm upon confirmation of rPD by BICR, TTCT was delayed for participants who had crossed over.
Time Frame: From date of randomization until date of subsequent chemotherapy or date of death from any cause, whichever comes first, assessed up to 43 months (estimated final OS analysis)
Reporting Status: Not Posted, anticipated posting 2026-09

10. Secondary Outcome: European Quality of Life (EuroQol) - 5 Domain 5 Level Scale (EQ-5D- 5L)
Description: EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. Higher scores indicated greater levels of problems across each of the five dimensions.
Time Frame: From randomization up till 30 day safety Follow-up or week 48 of long term Follow-up for patients prematurely discontinued, assessed up to 43 months
Reporting Status: Not Posted, anticipated posting 2026-09

11. Secondary Outcome: Functional Assessment of Cancer Therapy - Prostate (FACT-P) Questionnaire
Description: The FACT-P total score determines the level of prostate cancer specific health related quality of life (HRQoL). The higher the FACT-P score, the better the QoL. FACT-P assesses symptoms/problems related to prostate carcinoma and its treatment. It is a combination of the FACT- General + the Prostate Cancer Subscale (PCS). The FACTGeneral (FACT-G) is a 27 item Quality of Life (QoL) measure that provides a total score as well as subscale scores: Physical (0-28), Functional (0-28), Social (0-28), and Emotional Well-being (0-24). The total score range is between 1-108, higher scores indicates better for total score and subscale scores. PCS is a 12-item prostate cancer subscale that asks about symptoms and problems specific to prostate cancer (Range 0-48, higher scores better). The FACT-P total score is the sum of all 5 subscale scores of the FACT-P questionnaire and ranges from 0-156. Higher scores indicate higher degree of functioning and better quality of life.
Time Frame: as for outcome 10
Reporting Status: Not Posted, anticipated posting 2026-09

12. Secondary Outcome: Brief Pain Inventory - Short Form (BPI-SF) Questionnaire
Description: The BPI-SF is a publicly available instrument to assess the pain and includes severity and interference scores. BPI-SF is an 11-item selfreport questionnaire that is designed to assess the severity and impact of pain on daily functions of a participant. Pain severity score is a mean value for BPI-SF questions 3, 4, 5 and 6 (questions inquiring about the extent of pain, where the extent is ranked from 0 [no pain] to 10 [pain as bad as you can imagine]). Pain severity progression is defined as an increase in score of 30% or greater from baseline without decrease in analgesic use.
Time Frame: From screening up till 30 day safety Follow-up or week 48 of long term Follow-up for patients prematurely discontinued, assessed up to 43 months (estimated final OS analysis)
Reporting Status: Not Posted, anticipated posting 2026-09

13. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: The distribution of adverse events will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters. Treatment emergent adverse events falling into the category of myelosuppression, renal toxicity or second malignancy will be recorded beyond 30 day safety observation period.
Time Frame: From randomization till 30 day safety follow-up, assessed up to 43 months (estimated final OS analysis).
Reporting Status: Not Posted, anticipated posting 2026-09

ADVERSE EVENTS:
Time Frame: From start of study drug to max (30 days after EOT or last AAA617 dose date+41 days, last ARDT dose+30 days) or day before crossover up to data cut-off, max. of 42 months from randomization.
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up.
  The Safety Analysis Set was assessed for Serious and Other Adverse Events during the randomized On-Treatment Period.
Arm/Group | 177Lu-PSMA-617 | Androgen Receptor-directed Therapy (ARDT)
All-Cause Mortality (participants affected / at risk) | 142/234 | 157/234
Serious Adverse Events (participants affected / at risk) | 46/227 | 76/232
Other Adverse Events (participants affected / at risk) | 217/227 | 208/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 177Lu-PSMA-617 (N=227) | Androgen Receptor-directed Therapy (ARDT) (N=232)
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Aortic valve disease mixed (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Visual impairment (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 2
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Pain (General disorders) | 1 | 4
Polyp (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 3
COVID-19 pneumonia (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Infection (Infections and infestations) | 1 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 3
Pyelonephritis (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 0
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 4
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 3
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 3
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Coma (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Meningism (Nervous system disorders) | 1 | 0
Neurotoxicity (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 1
Spinal cord compression (Nervous system disorders) | 1 | 5
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 5
Haematuria (Renal and urinary disorders) | 0 | 3
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Renal haemorrhage (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 3
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Urine abnormality (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 177Lu-PSMA-617 (N=227) | Androgen Receptor-directed Therapy (ARDT) (N=232)
Anaemia (Blood and lymphatic system disorders) | 59 | 44
Neutropenia (Blood and lymphatic system disorders) | 12 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 17 | 7
Dry eye (Eye disorders) | 14 | 2
Constipation (Gastrointestinal disorders) | 49 | 32
Diarrhoea (Gastrointestinal disorders) | 38 | 23
Dry mouth (Gastrointestinal disorders) | 135 | 6
Nausea (Gastrointestinal disorders) | 73 | 29
Vomiting (Gastrointestinal disorders) | 26 | 12
Asthenia (General disorders) | 72 | 66
Fatigue (General disorders) | 54 | 59
Oedema peripheral (General disorders) | 19 | 29
Pain (General disorders) | 6 | 12
COVID-19 (Infections and infestations) | 36 | 26
Fall (Injury, poisoning and procedural complications) | 6 | 14
Blood alkaline phosphatase increased (Investigations) | 14 | 18
Lymphocyte count decreased (Investigations) | 12 | 3
Weight decreased (Investigations) | 15 | 32
Decreased appetite (Metabolism and nutrition disorders) | 49 | 44
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 46 | 54
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 45
Bone pain (Musculoskeletal and connective tissue disorders) | 20 | 17
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 10 | 16
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 | 27
Dizziness (Nervous system disorders) | 11 | 13
Dysgeusia (Nervous system disorders) | 19 | 6
Headache (Nervous system disorders) | 19 | 11
Insomnia (Psychiatric disorders) | 8 | 13
Haematuria (Renal and urinary disorders) | 4 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Hot flush (Vascular disorders) | 15 | 22
Hypertension (Vascular disorders) | 6 | 22

LIMITATIONS AND CAVEATS:
235 participants were randomized to the AAA617 arm and 234 to the ARDT arm. However, only 228 participants in the AAA617 arm and 232 in the ARDT arm received at least one dose of study treatment. Additionally, 1 participant in the AAA617 arm was excluded from the safety analysis set due to a protocol violation, which means only 227 participants were included in the safety analysis set for this arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT04689828/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT04689828/SAP_001.pdf